CLINICAL TRIAL: NCT00068900
Title: FFA Metabolism in Different Types of Human Obesity
Status: Withdrawn | Type: Observational
Why Stopped: NOT A CLINICAL TRIAL
Sponsor: Mayo Clinic (Other)
Other Study IDs: FFAMET - dk40484 (withdrawn)
Record Dates: First submitted 2003-09-10; First posted 2003-09-12 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
We will give intravenous fat molecules to help us understand how the fat that is released from peoples fat cells is used. This will be done when people are eating, not eating and walking.

ELIGIBILITY:
Inclusion Criteria: BMI 28-36 -upper body obesity and lower body obesity non-obese BMI 19-24. Females premenopausal. Must be a non-smoker.

Exclusion Criteria: BP> 160/95 on HTN meds, known systemic illness. Medications that affect fat metabolism. We do no cover travel expenses. Known heart and vascular disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2003-11; Primary Completion 2004-01 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States